CLINICAL TRIAL: NCT00175955
Title: An 8-week Exploratory, Double-blind, Placebo Controlled, Randomized Trial: Evaluation of the Efficacy and Safety of Levetiracetam up to 3000 mg/Day (250-500 mg Oral Tablets in b.i.d. Administration) on Neuroleptic-induced Tardive Dyskinesia in Subjects With Stable Axis I Psychiatric Disorder, Aged From at Least 18 Years to 80 Years.
Brief Title: Levetiracetam in the Treatment of Neuroleptic-induced Tardive Dyskinesia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: UCB Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: N01142; EudraCT Number 2004-001302-27
Record Dates: First submitted 2005-09-09; First posted 2005-09-15 (Estimated); Last update posted 2013-12-06 (Estimated); Status verified 2009-09

CONDITIONS: Dyskinesia, Medication-induced
Keywords: Neuroleptic-induced tardive dyskinesia; Keppra, Levetiracetam
MeSH Terms: conditions — Dyskinesia, Drug-Induced | interventions — Levetiracetam

INTERVENTIONS:
Drug: Levetiracetam

SUMMARY:
An 8-week study to examine safety and efficacy of levetiracetam in patients with neuroleptic-induced tardive dyskinesia

ELIGIBILITY:
Inclusion Criteria:

* Subjects between ages 18 and 80 years
* Subjects must have a diagnosis of stable axis I psychiatric disorder at least 6 months prior to screening
* Subjects must have a stable neuroleptic-induced tardive dyskinesia at least 1 month prior to screening and meet tardive dyskinesia severity criteria
* Subjects must have used antipsychotics for at least 6 cumulative months, and, be on a stable dose for 1 month prior to screening

Exclusion Criteria:

* Presence of any axis II condition within 6 months prior to screening
* Huntington´s disease, idiopathic dystonia, Wilson´s disease, Sydenham´s chorea, thyroid dysfunction, spontaneous dyskinesia
* Start of drugs-other than neuroleptics- that can cause dyskinesia
* Presence of additional major disease such as cardiac, renal or hepatic dysfunction or terminal illness

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 70
Dates: Start 2005-05; Primary Completion 2005-12 (Actual); Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
Reduction in neuroleptic-induced tardive dyskinesia over an 8 week treatment period

SECONDARY OUTCOMES:
Neuroleptic-induced akathisia and other extrapyramidal symptoms ,
Effect on the primary psychiatric disorder
Safety

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — UCB Pharma
Locations (7):
- Belgium (6):
  - Antwerp
  - Bourgois
  - Gonce
  - Hulselmans
  - Liège
  - Roeselare
- Haralanov, Bulgaria